CLINICAL TRIAL: NCT02593773
Title: Multicenter, Safety and Efficacy, Open-Label Extension Study of ACTIMMUNE® (Interferon γ-1b) in Children and Young Adults With Friedreich's Ataxia
Brief Title: Safety, Tolerability and Efficacy of ACTIMMUNE® Dose Escalation in Friedreich's Ataxia Study
Acronym: STEADFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-ACT-302
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Friedreich's Ataxia
Keywords: Interferon gamma
MeSH Terms: conditions — Friedreich Ataxia | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- interferon γ-1b (Experimental): Subcutaneous (SC) doses of ACTIMMUNE® TIW for a total of 26 weeks.
  Interventions: Drug: Interferon γ-1b

INTERVENTIONS:
Drug: Interferon γ-1b — The study drug dose is planned to be escalated on a weekly basis over the first 4 weeks of treatment (from 10 µg/m² to 25, 50, and 100 µg/m²). The dose may be reduced, interrupted, or held based on tolerability. By Week 13, all participants are to be on a stable tolerated dose of study drug in order to continue study participation; the dose may not be further increased after Week 13, however, it may be reduced on a case-by-case basis to manage drug-related adverse events (AEs).
  Other Names: ACTIMMUNE®

SUMMARY:
The purpose of this phase 3 multi-center, open-label extension study is to evaluate the long-term safety of ACTIMMUNE® (interferon-γ 1b) in participants with Friedreich's Ataxia.

DETAILED DESCRIPTION:
Participants who complete 26 weeks of blinded treatment in HZNP-ACT-301 (NCT02415127), will be eligible to enter this 6-month study. All participants will receive ACTIMMUNE® 3 times a week (TIW) for 26 weeks. In order to maintain the study blind in HZNP-ACT-301 (NCT02415127), all participants in this open-label extension study will undergo ACTIMMUNE® titration, regardless if they received ACTIMMUNE® or placebo in HZNP-ACT-301 (NCT02415127). The Week 26 Visit from HZNP-ACT-301 (NCT02415127) will serve as the Baseline Visit (Day 1) for this study. During the treatment period, additional clinic visits are scheduled at Weeks 4, 13, and 26; in between clinic visits, participants (and/or caregivers) will be monitored via emails/phone calls on a weekly basis until participants reach their maximum tolerated dose, and on a monthly basis thereafter.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and child assent, if applicable.
* Completed 26 weeks of blinded treatment in Study HZNP-ACT-301 (NCT02415127).
* If female, the subject is not pregnant or lactating or intending to become pregnant during the study, or within 30 days after the last dose of study drug. Female subjects of child-bearing potential must have a negative urine pregnancy test result at Baseline/Day 1 (Week 26 of Study HZNP-ACT-301 [NCT02415127]), and agree to use a reliable method of contraception throughout the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* Subjects will be ineligible if, in the opinion of the Investigator, they are unlikely to comply with the study protocol or have a concomitant disease or condition that could interfere with the conduct of the study or potentially put the subject at unacceptable risk.

NOTE: Additional inclusion/exclusion criteria may apply.

Ages: 10 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2015-12-25 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - University of California, Los Angeles Neurology Clinic, Los Angeles, California
  - University of Florida - Clinical Research Center, Gainesville, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon γ-1b: Subcutaneous (SC) ACTIMMUNE® 3 times a week (TIW) for a total of 26 weeks. The study drug dose was escalated on a weekly basis over the first 4 weeks of treatment (from 10 μg/m² to 25, 50, and 100 μg/m²), based on tolerability, with all participants on a stable tolerated dose by Week 13. Dose may have been reduced, interrupted, or held based on tolerability thereafter.
Period: Overall Study
Arm/Group | Interferon γ-1b
Started | 86
Completed | 51
Not Completed | 35
Not completed — Voluntary Withdrawal | 3
Not completed — Study Terminated by Sponsor | 31
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Interferon γ-1b: SC ACTIMMUNE® TIW for a total of 26 weeks. The study drug dose was escalated on a weekly basis over the first 4 weeks of treatment (from 10 μg/m² to 25, 50, and 100 μg/m²), based on tolerability, with all participants on a stable tolerated dose by Week 13. Dose may have been reduced, interrupted, or held based on tolerability thereafter.
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (4.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 81
  More than one race | 2
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: An adverse event (AE) is any untoward medical occurrence, whether or not the event is considered related to the investigational product. A TEAE is any adverse change from the subject's baseline condition, including any laboratory test value abnormality judged as clinically significant by the investigator, that occurs on or after the date of the first dose of study drug administered at home and throughout the duration of the clinical study, whether the adverse event is considered related to the treatment or not. An SAE is an AE that results in death, is life-threatening, results in persistent or significant disability or incapacity, inpatient hospitalization or prolongation of an existing hospitalization, is a congenital anomaly or birth defect, or other medically important event.
Time Frame: Baseline/Day 1 (Week 26 of Study HZNP-ACT-301 [NCT02415127]) through Week 28 (follow-up safety visit)
Population: Safety Population, defined as all participants who received at least 1 dose of open-label study drug after the Baseline Visit.
Measure: Number; unit: participants
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 86
participants
  ≥ 1 TEAE | 78
  ≥ 1 Related TEAE | 61
  ≥ 1 SAE | 4
  ≥ 1 Related SAE | 0
  ≥ 1 TEAE Leading to Discontinuation | 1
  ≥ 1 TEAE Leading to Death | 1

2. Primary Outcome: Number of Participants With Positive/Negative Neutralizing Antibody (NAb) and Anti-Drug Antibody (ADA) Tests
Description: NAb testing only for those participants with a positive ADA test. Baseline is defined as the last non-missing measurement/assessment on the date of Week 26 Visit from study HZNP-ACT-301 (NCT02415127). If this measurement was missing or otherwise unavailable, it was the last non-missing measurement/assessment on or prior to first dose in this study. If the participant discontinued the study, then premature withdrawal assessments were mapped to the nearest scheduled visit based on schedule of the assessment and the study day. If the mapped visit was already available then the visit was mapped to the next schedule visit. Last on study assessment is the last non-missing post-baseline assessment for each participant.
Time Frame: Baseline/Day 1 (Week 26 of Study HZNP-ACT-301 [NCT02415127]), Week 4, Week 13, Week 26, and Week 28 (follow-up safety visit)
Population: Safety Population, defined as all participants who received at least 1 dose of open-label study drug after the Baseline Visit. Participants with an assessment at each time point are presented.
Measure: Number; unit: participants
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 86
participants
  Baseline ADA = negative | 85
  Baseline ADA = positive | 1
  Baseline NAb = negative: number analyzed (Participants) | 1
  Baseline NAb = negative | 1
  Baseline NAb = positive: number analyzed (Participants) | 1
  Baseline NAb = positive | 0
  Week 4 ADA = negative: number analyzed (Participants) | 84
  Week 4 ADA = negative | 84
  Week 4 ADA = positive: number analyzed (Participants) | 84
  Week 4 ADA = positive | 0
  Week 4 NAb = negative: number analyzed (Participants) | 0
  Week 4 NAb = positive: number analyzed (Participants) | 0
  Week 13 ADA = negative: number analyzed (Participants) | 79
  Week 13 ADA = negative | 79
  Week 13 ADA = positive: number analyzed (Participants) | 79
  Week 13 ADA = positive | 0
  Week 13 NAb = negative: number analyzed (Participants) | 0
  Week 13 NAb = positive: number analyzed (Participants) | 0
  Week 26 ADA = negative: number analyzed (Participants) | 64
  Week 26 ADA = negative | 64
  Week 26 ADA = positive: number analyzed (Participants) | 64
  Week 26 ADA = positive | 0
  Week 26 NAb = negative: number analyzed (Participants) | 0
  Week 26 NAb = positive: number analyzed (Participants) | 0
  Week 28 (Follow-up) ADA = negative: number analyzed (Participants) | 56
  Week 28 (Follow-up) ADA = negative | 56
  Week 28 (Follow-up) ADA = positive: number analyzed (Participants) | 56
  Week 28 (Follow-up) ADA = positive | 0
  Week 28 (Follow-up) NAb = negative: number analyzed (Participants) | 0
  Week 28 (Follow-up) NAb = positive: number analyzed (Participants) | 0
  Last On Study Assessment ADA = negative: number analyzed (Participants) | 85
  Last On Study Assessment ADA = negative | 85
  Last On Study Assessment ADA = positive: number analyzed (Participants) | 85
  Last On Study Assessment ADA = positive | 0
  Last On Study Assessment NAb = negative: number analyzed (Participants) | 0
  Last On Study Assessment NAb = positive: number analyzed (Participants) | 0

3. Primary Outcome: Change From Baseline to Week 26 in the Friedreich's Ataxia Rating Scale (FARS)-mNeuro Score
Description: The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions were assessed. The FARS-mNeuro score excludes the peripheral nervous system subscale score and the facial and tongue atrophy and fasciculations from the bulbar subscale score. Scores range from 0 (normal) to 93 (most impairment). A negative change from baseline is an improvement.
Time Frame: From Baseline to Week 26 for all participants and from Baseline of HZNP-ACT-301 (NCT02415127)to Week 26 of HZNP-ACT-302 (52-week treatment duration) for participants receiving active treatment in both studies.
Population: Because the Sponsor discontinued the development of ACTIMMUNE® for the treatment of Friedreich's Ataxia, the planned analyses of the efficacy endpoints were not conducted. Any raw data collected for this endpoint exist as by-subject listings only, and are unanalyzed per protocol.
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline to Week 26 in Activities of Daily Living (ADL) Score
Description: Participants and/or their caregivers rated 9 areas of daily living skills (speech, swallowing, cutting food and handling utensils, dressing, personal hygiene, falling, walking, quality of sitting position, and bladder function) on a 5-point scale (0=normal, 4=greatest loss of function) with allowable increments of 0.5 if the participant or caregiver strongly felt that a task falls between 2 scores. ADL scores can range from 0 (normal) to 36 (greatest loss of function). A negative change from baseline indicates improvement.
Time Frame: as for outcome 3
Population: as for outcome 3
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline at Week 26 in Timed 25-Foot Walk (T25FW)
Description: The T25FW is a quantitative measure of lower extremity function. Participants are directed to 1 end of a clearly marked 25-foot course and instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the participant walk back the same distance, and the score for the test is the average of the 2 walks (after reciprocal transformation). Participants may use assistive devices when performing this task, with the same assistive device used at each assessment. A negative change from Baseline indicates improvement.
Time Frame: as for outcome 3
Population: as for outcome 3
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of FARS-mNeuro Responders and Non-Responders at Week 26
Description: A participant was considered a responder if they had an improvement (decrease) of at least 3 points from Baseline at Week 26 for the FARS-mNeuro score. The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions were assessed. The FARS-mNeuro score excludes the peripheral nervous system subscale score and the facial and tongue atrophy and fasciculations from the bulbar subscale score. Scores range from 0 (normal) to 93 (most impairment).
Time Frame: Week 26
Population: as for outcome 3
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline to Week 26 in Total Friedreich Ataxia Rating Scale Score (FARStot)
Description: The FARS assessment includes neurological signs that specifically reflect neural substrates affected in FA. Based on a neurological examination, bulbar, upper limb, lower limb, peripheral nerve, and upright stability/gait functions are assessed. FARStot scores range from 0 (normal) to 125 (most impairment). A negative change from baseline indicates improvement.
Time Frame: as for outcome 3
Population: as for outcome 3
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Post-dose on Day 1 (Week 26 of Study HZNP-ACT-301 [NCT02415127]) through Week 28 (follow-up safety visit) for Serious TEAEs, and through the end of the study (Week 26) for nonserious TEAEs.
Arm/Group | Interferon γ-1b
All-Cause Mortality (participants affected / at risk) | 1/86
Serious Adverse Events (participants affected / at risk) | 4/86
Other Adverse Events (participants affected / at risk) | 66/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon γ-1b (N=86)
Atrial fibrillation (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Eosinophilic myocarditis (Cardiac disorders) | 1
Chest pain (General disorders) | 2
Sepsis (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Heart rate increased (Investigations) | 1
Haemodynamic instability (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon γ-1b (N=86)
Neutropenia (Blood and lymphatic system disorders) | 18
Abdominal pain upper (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 13
Chills (General disorders) | 5
Fatigue (General disorders) | 7
Pain (General disorders) | 7
Pyrexia (General disorders) | 15
Gastroenteritis viral (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 7

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the development of ACTIMMUNE® for the treatment of Friedreich's Ataxia was discontinued after Study HZNP-ACT-301 (NCT02415127) failed to meet its primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .

DOCUMENTS (2):
  • Study Protocol (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT02593773/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT02593773/SAP_001.pdf